CLINICAL TRIAL: NCT01827579
Title: Adoptive Immunotherapy With CD25/71 Allodepleted Donor T Cells to Improve Immunity After Unrelated Donor Stem Cell Transplant
Brief Title: Infusion of Depleted T Cells Following Unrelated Donor Stem Cell Transplant (ICAT)
Acronym: ICAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCL/11/0519; 2013-000872-14 (EudraCT Number); MR/K007491/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Haematological Malignancies
Keywords: Transplant; CD25/71 allodepleted donor T cells; Infection; Acute Myeloid Leukaemia; Acute Lymphoblastic Leukaemia; Adult; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Infections; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD25/71 allodepleted donor T-cells (Experimental): CD25/71 allodepleted donor T-cells will be administered at a dose of 10^5 /kg at day 30 post-SCT, 3 x 10^5 /kg at day 60 and 10^6 /kg at day 90 post transplant
  Interventions: Biological: CD25/71 allodepleted donor T-cells
- Control (normal HSCT) (No Intervention): Patients randomised to the control arm with undergo stem cell transplantation according to site local practice.

INTERVENTIONS:
Biological: CD25/71 allodepleted donor T-cells — CD25/71 allodepleted donor T-cells will be administered at a dose of 10^5 /kg at day 30 post-SCT, 3 x 10^5 /kg at day 60 and 10^6 /kg at day 90 post transplant
  Arms: CD25/71 allodepleted donor T-cells

SUMMARY:
The purpose of this study is to evaluate whether the administration of allodepleted donor T cells to patients with haematological malignancies after stem cell transplant can improve the recovery of the patients immune system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* Underlying haematological malignancy
* Planned allogeneic peripheral blood stem cell transplantation from a 10/10 or 9/10 HLA matched unrelated donor, using an Alemtuzumab-based conditioning protocol
* Written Informed consent

Exclusion Criteria:

* Life expectancy < 6 weeks
* Female patients who are pregnant and lactating
* Patients who are serologically positive for Hepatitis B, C or HIV pre-SCT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Circulating CD3+ve T cell count at 4 months post-SCT | 4 months post transplant

SECONDARY OUTCOMES:
Incidence of grade II-IV acute and chronic GVHD | 1 year post transplant
Time to recovery of normal T-cell (>700/uL) and CD4 (>300/uL) counts and normal TCR diversity as assessed by Vb spectratyping | 1 year post transplant
In vitro anti-viral responses of circulating PBMC | 1 year post transplant
Transplant related mortality at 1 year post-SCT | 1 year post transplant
Disease-free survival at 1 year post-SCT | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Persis Amrolia, Study Chair — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University College London Hospital, London
  - Manchester Royal Infirmary, Manchester